CLINICAL TRIAL: NCT00042562
Title: Open-Label Treatment With Duloxetine Hydrochloride Once-Daily Dosing for Evaluation of Stabilization Dose in Patients With Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6476; F1J-US-HMBZ
Record Dates: First submitted 2002-07-31; First posted 2002-08-05 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Major Depressive Disorder
Keywords: Depressed; blues; sadness; feelings of guilt; hopelessness; lack of energy
MeSH Terms: conditions — Depressive Disorder, Major; Consciousness Disorders; Fatigue | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine

SUMMARY:
The purposes of this study are to determine:

The safety of duloxetine and any side effects that might be associated with it.

Whether duloxetine can help patients with major depression.

The safety associated with switching from a medication you may be taking for depression to taking duloxetine.

It is possible that information collected during this study will be analyzed by the sponsor in the future to evaluate duloxetine for other possible uses or for other medical or scientific purposes other than those currently proposed.

ELIGIBILITY:
Inclusion Criteria:

* You must be at least 18 years old.
* You must have been diagnosed with major depressive disorder.
* You must be able to visit the doctor's office once a week to once every 2 weeks for a total of 14 weeks

Exclusion Criteria:

* You are a woman and are pregnant or breastfeeding.
* You have a current or previous major psychiatric disorder other than depression, such as bipolar disorder, schizophrenia, or other psychotic disorder.
* You have had a primary diagnosis of an anxiety disorder within the past 6 months.
* You have a history of alcohol or drug dependence or abuse within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Carlsbad, California
  - Los Angeles, California
  - Stanford, California
  - Cromwell, Connecticut
  - Coral Springs, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Bangor, Maine
  - Boston, Massachusetts
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - West Allis, Wisconsin